CLINICAL TRIAL: NCT00111787
Title: A Phase II Study to Evaluate the Efficacy, Safety, and Pharmacodynamics of Lapatinib in Combination With Paclitaxel as Neoadjuvant Therapy in Patients With Newly Diagnosed Inflammatory Breast Cancer
Brief Title: Study Of Lapatinib In Combination With Paclitaxel In The Treatment Of Newly Diagnosed Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF102580
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms, Breast
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall study (Experimental): A Single arm study with 2 cohorts of participants. Cohort A consists of participants with tumors overexpressing HER2 and/or EGFR. Cohort B consists of participants with tumors expressing EGFR without overexpressing HER2.
  Interventions: Drug: Lapatinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Lapatinib — Daily-monotherapy [1500 milligrams (mg)] for 14 days, then daily combination therapy (with weekly paclitaxel) for 12 weeks
Drug: Paclitaxel — Weekly (80mg/m^2) combination therapy (with daily Lapatinib) for 12 weeks
  Other Names: Lapatinib

SUMMARY:
This Study was designed to determine how effective and safe a new investigational drug, lapatinib, is in combination with paclitaxel in treating patients with newly diagnosed inflammatory breast cancer. Tumor tissue collected pre-treatment, following 14 days of treatment and at the time of surgical resection will be examined for pathologic response and biologic activity by IHC (immunohistochemistry) within the tumor. Treatment will consist of 14 days of lapatinib monotherapy followed by 12 weeks of combination therapy with lapatinib and paclitaxel. Blood samples for hematology and chemistry panels, MUGA/ECHO exams and physical exams will be performed throughout the study to monitor safety.

ELIGIBILITY:
Inclusion criteria:

* Tumor accessible for multiple biopsies
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Adequate bone marrow
* Renal and hepatic function
* LVEF (left ventricular ejection fraction) greater than 0% based on ECHO (echocardiogram) or MUGA (multigated acquisition).

Exclusion criteria:

* Females who are pregnant or nursing.
* Any unstable, pre-existing major medical condition.
* Received an investigational drug within the past 4 weeks.
* Had major surgery in the past 2 weeks.
* Currently receiving amiodarone or has received amiodarone in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-04-11 (Actual); Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with pathologic complete response rate (pCR) | Week 12
  pCR was defined as the percentage of participants who achieved an assessment of complete response (CR) following pathologic review of resected tissue. CR was the disappearance of all target lesions. Participants in each cohort with unknown or missing response (i.e., those that did not undergo surgery) were included in the denominator when calculating the percentage. From an efficacy standpoint, the HER2+ population response was considered to be of special interest.

SECONDARY OUTCOMES:
Percentage of participants with pCR that underwent surgical resection | Week 12
  pCR for participants that underwent surgical (surg) resection was defined as the percentage of participants within each cohort who achieved an assessment of CR following pathologic review of resected tissue. CR was the disappearance of all target lesions. Participants in each cohort that did not undergo surgical resection were excluded from the denominator when calculating the percentage. From an efficacy standpoint, the HER2+ population response was considered to be of special interest.
Percentage of participants with objective response rate (ORR) at the end of study (Response evaluation criteria in solid tumor [RECIST]) | Week 14
  ORR at the end of the study was defined as the number of participants within each cohort who had a confirmed CR or partial response (PR) at the end of the study divided by the total number of participants enrolled in each cohort. CR was the disappearance of all target lesions. PR was at least a 30 percent decrease in the sum of the longest diameter of target lesions, taking as a reference, the Baseline sum longest diameter. Each participant's response was based on the investigator assessment of best response using RECIST criteria. Participants in each cohort with unknown or missing response was treated as non-responders; i.e. they were included in the denominator when calculating the percentage. From an efficacy standpoint, the HER2+ population was considered to be of special interest.
Percentage of participants with ORR at the end of study (Clinically Evaluable Skin Disease Criteria) | Week 14
  ORR at the end of the study was defined as the number of participants within each cohort who had a confirmed CR or PR at the end of the study divided by the total number of participants enrolled in each cohort. CR was the disappearance of all target lesions. PR was at least a 30 percent decrease in the sum of the longest diameter of target lesions, taking as a reference, the Baseline sum longest diameter. Each participant's response was based on the investigator assessment of best response using Clinically Evaluable Skin Disease Criteria. Participants in each cohort with unknown or missing response was treated as non-responders; i.e. they were included in the denominator when calculating the percentage. From an efficacy standpoint, HER2+ population was considered to be of special interest.
Percentage of participants with ORR at the end of study ('Best' of RECIST and Clinically Evaluable Skin Disease Criteria) | Week 14
  ORR at the end of the study was defined as the number of participants within each cohort who had a confirmed CR or PR at the end of the study divided by the total number of participants enrolled in each cohort. CR was the disappearance of all target lesions. PR was at least a 30 percent decrease in the sum of the longest diameter of target lesions, taking as a reference, the Baseline sum longest diameter. The best response of the participant was defined by the 'Best' combined response (RECIST and Clinically Evaluable Skin Disease Criteria) provided there is no evidence of disease progression. Participants in each cohort with unknown or missing response was treated as non-responders; i.e. they were included in the denominator when calculating the percentage. From an efficacy standpoint, the HER2+ population was considered to be special interest.
Percentage of participants with investigator-Assessed Best Response at the end of monotherapy phase (Day 14) (Clinically Evaluable Skin Disease Criteria) | Day 14
  ORR at the end of the monotherapy phase was defined as the percentage of participants within each cohort who had a confirmed CR or PR at the end of lapatinib monotherapy (Day 14) divided by the total number of participants enrolled in each cohort. CR was the disappearance of all target lesions. PR was at least a 30 percent decrease in the sum of the longest diameter of target lesions, taking as a reference, the Baseline sum longest diameter. Each participant's response was based on the investigator assessment of best response using clinically evaluable skin disease criteria. Participants in each cohort with unknown or missing response was treated as non-responders; i.e. they were included in the denominator when calculating the percentage. From an efficacy standpoint, the HER2+ population was considered to be special interest.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Week 14, surgical resection and post treatment
  An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE was defined as any untoward medical occurrence that, at any dose that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect, resulted in deterioration in left ventricular cardiac function and caused Grade 3 or 4 interstitial pneumonitis.
Number of participants with shift from Baseline in hematological toxicity grade | Day 14 and up to Week 23, surg resection and post treatment
  Hematology was summarized for hemoglobin (Hb), platelets, white blood cell count (WBC), neutrophils (Neu), lymphocytes by scheduled assessment and also according to the maximum common terminology criteria (CTC) toxicity grade. Baseline was the most recent lab value prior to and within two weeks of the first dose of lapatinib. Change from Baseline was calculated as the value at each visit minus Baseline value.
Number of participants with shift from Baseline in clinical chemistry toxicity grade | Day 14, Week 4, 8, 12, 16, 20, Surg resection and post treatment
  Clinical chemistry was summarized for sodium, potassium (K), bicarbonate (bicarb), albumin (alb), calcium, gamma glutamyl transferase (GGT), creatinine (creat), total bilirubin (TB), alkaline phosphatase (ALP), aspartate amino transferase (AST) and alanine amino transferase (ALT) by scheduled assessment and also according to the maximum CTC toxicity grade. Baseline was the most recent lab value prior to and within two weeks of the first dose of lapatinib. Change from Baseline was calculated as the value at each visit minus Baseline value.
Change from Baseline in vital signs- Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) | Day 14, Week 1 and up to Week 24, surg resection and post treatment
  Vitals signs (SBP and DBP) were assessed from screening until the post treatment phase. Baseline was the most recent blood pressure (BP) mean prior to the first dose of lapatinib. Change from Baseline was calculated as the mean at each visit minus the mean at Baseline.
Change from Baseline in vital signs- Heart Rate (HR) | Day 14, Week 1 and up to Week 24, surg resection and post treatment
  Vitals signs (HR) were assessed from screening until the post treatment phase. Baseline was the most recent BP mean prior to the first dose of lapatinib. Change from Baseline was calculated as the mean at each visit minus the mean at Baseline.
Change from Baseline in vital signs- Body temperature | Day 14, Week 1 and up to Week 24, surg resection and post treatment
  Vitals signs (body temperature) were assessed from screening until the post treatment phase. Baseline was the most recent BP mean prior to the first dose of lapatinib. Change from Baseline was calculated as the mean at each visit minus the mean at Baseline.
Number of participants with abnormal electrocardiogram (ECG) findings | Screening and unscheduled
  ECG was performed at screening and at unscheduled visits. Participants with abnormal clinically significant and abnormal not clinically significant ECG findings was reported.
Number of participants with change from Baseline in echocardiogram (ECHO) or Multi-gated angiogram (MUGA) results at any post Baseline visit | Screening, Week 8, 16, 24, post treatment
  For ECHO and MUGA scans, the left ventricular ejection fraction (percent) was summarized for each scheduled assessment. Absolute change from Baseline was summarized according to the following categories: any increase, 0 to less than 20 percent decrease, >=20 percent decrease or >=20 percent decrease and below the lower limit of normal (LLN). Baseline was the most recent ECOG evaluation prior to the first dose of lapatinib. Change from Baseline was calculated as the value at the post treatment minus Baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (4):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Zion, Illinois
  - GSK Investigational Site, Houston, Texas
- Australia (7):
  - GSK Investigational Site, Campbelltown, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
- GSK Investigational Site, Toronto, Ontario, Canada
- France (3):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
- GSK Investigational Site, Ramat Gan, Israel
- GSK Investigational Site, Auckland, New Zealand
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Valencia
- Tunisia (2):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Tunis
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Background] Boussen H, Cristofanilli M, Zaks T, DeSilvio M, Salazar V, Spector N. Phase II study to evaluate the efficacy and safety of neoadjuvant lapatinib plus paclitaxel in patients with inflammatory breast cancer. J Clin Oncol. 2010 Jul 10;28(20):3248-55. doi: 10.1200/JCO.2009.21.8594. Epub 2010 Jun 7. PMID 20530274